CLINICAL TRIAL: NCT03423797
Title: Effectiveness of Biannual Application of Silver Nitrate Solution Followed by Sodium Fluoride Varnish With or Without Functionalized Tricalcium Phosphate in Arresting Caries in Preschool Children
Brief Title: The Caries-arresting Effect of Incorporating fTCP to NaF Varnish Applied Following AgNO3 in Preschool Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chun-Hung Chu, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 17-176
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Early Childhood Caries
Keywords: silver nitrate; sodium fluoride; dental caries; equivalence trial
MeSH Terms: conditions — Dental Caries | interventions — 4-fluoro-1-(1-(2-thienyl)cyclohexyl)piperidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NaF without fTCP (Active Comparator): 25% AgNO3 solution followed by 5% NaF.
  Interventions: Drug: 25% AgNO3 solution followed by 5% NaF
- NaF with fTCP (Experimental): 25% AgNO3 solution followed by 5% NaF with fTCP.
  Interventions: Drug: 25% AgNO3 solution followed by 5% NaF with fTCP

INTERVENTIONS:
Drug: 25% AgNO3 solution followed by 5% NaF — Dosage: 25% AgNO3 solution 7.9mg(Ag+)/0.05ml (max dose), 5% NaF: 11.6mg (F-)/0.5ml (max dose).
  Other Names: 5% NaF without fTCP
  Arms: NaF without fTCP
Drug: 25% AgNO3 solution followed by 5% NaF with fTCP — Dosage: 25% AgNO3 solution 7.9mg(Ag+)/0.05ml (max dose), 5% NaF with fTCP: 11.6mg (F-)/0.5ml (max dose).
  Other Names: 5% NaF with fTCP
  Arms: NaF with fTCP

SUMMARY:
The objective of this study is to compare the effectiveness of 25% AgNO3 solution plus 5% NaF varnish and 25% AgNO3 solution plus 5% NaF varnish with fTCP when applied semi-annually over 30 months in arresting dentine caries of primary teeth among preschool children. Half of Participants will receive topical application of 25% AgNO3 solution and 5% NaF varnish, while the other half will receive topical application of 25% AgNO3 solution and 5% NaF varnish with fTCP.

DETAILED DESCRIPTION:
Aim:The objective of this study is to compare the effectiveness of commercially available of 25% AgNO3 solution plus 5% NaF varnish and 25% AgNO3 solution plus 5% NaF varnish with fTCP when applied semi-annually over 30 months in arresting dentine caries of primary teeth among preschool children.

Methods: The extension of the Consolidated Standards of Reporting Trials 2010 Statement will be followed for this 30-month, randomised, double-blinded, equivalence clinical trial. Approximately 2,000 kindergarten children will be screened and at least 376 children with caries will be recruited. This sample size is sufficient for an appropriate statistical analysis. The children will be randomly allocated into 2 groups to treat their caries over a 30-month period: Group A - biannual application of a 25% AgNO3 solution followed by a 5% NaF varnish, and Group B - biannual application of a 25% AgNO3 solution followed by a 5% NaF varnish with functionalized tricalcium phosphate (fTCP).Clinical examinations will be conducted at 6-month intervals to assess whether the caries are arrested (primary outcome). Confounding factors such as oral hygiene habits will be collected through a parental questionnaire.

Possible results and implications: As the first of its kind, this study would help to determine whether AgNO3 followed by 5% NaF varnish with and without fTCP are equivalent in arresting dentine caries of primary teeth in preschool children when applied semi-annually.

ELIGIBILITY:
Inclusion Criteria:

* have at least one tooth with cavitated dentine carious lesion

Exclusion Criteria:

* Children have severe forms of dental hypoplasia, under dental treatment or wearing orthodontic devices, have major systemic illness, and are on long-term medication.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 408 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
The hardness of cavity on tooth by probing | The follow-up oral examinations will be conducted every 6 months for 30 months totally
  The effectiveness of adjunctive application of 25% AgNO3 solution and 5% NaF varnish with or without fTCP is expected to be equivalent in arresting dentine caries of primary teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Chun Hung Chu, Ph.D, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Chen KJ, Gao SS, Duangthip D, Lo ECM, Chu CH. Randomized Clinical Trial on Sodium Fluoride with Tricalcium Phosphate. J Dent Res. 2021 Jan;100(1):66-73. doi: 10.1177/0022034520952031. Epub 2020 Aug 31. PMID 32866050
- [Derived] Chen KJ, Gao SS, Duangthip D, Lo ECM, Chu CH. The caries-arresting effect of incorporating functionalized tricalcium phosphate into fluoride varnish applied following application of silver nitrate solution in preschool children: study protocol for a randomized, double-blind clinical trial. Trials. 2018 Jul 4;19(1):352. doi: 10.1186/s13063-018-2741-1. PMID 29973256